CLINICAL TRIAL: NCT01543152
Title: A Phase I, Open-Label Study to Assess the Effect of Escalating Doses of Cyclophosphamide on the Engraftment of SB-728-T in Aviremic HIV-Infected Subjects on HAART
Brief Title: Dose Escalation Study of Cyclophosphamide in HIV-Infected Subjects on HAART Receiving SB-728-T
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-728-1101
Record Dates: First submitted 2012-03-01; First posted 2012-03-02 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: HIV; autologous cell therapy; cyclophosphamide
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 - IV cyclophosphamide 200 mg (Experimental)
  Interventions: Genetic: SB-728-T
- Cohort 2 - IV cyclophosphamide 0.5 g/m2 (Experimental)
  Interventions: Genetic: SB-728-T
- Cohort 3 - IV cyclophosphamide 1.0 g/m2 (Experimental)
  Interventions: Genetic: SB-728-T
- Cohort 4 - IV cyclophosphamide 2.0 g/m2 (Experimental)
  Interventions: Genetic: SB-728-T
- Cohort 5 - IV cyclophosphamide 1.5 g/m2 (Experimental)
  Interventions: Genetic: SB-728-T

INTERVENTIONS:
Genetic: SB-728-T — Infusion will be 5 to 30 billion ZFN modified CD4+ T cells 1 day following IV cyclophosphamide 200 mg
  Other Names: cyclophosphamide
  Arms: Cohort 1 - IV cyclophosphamide 200 mg
Genetic: SB-728-T — Infusion will be 5 to 30 billion ZFN modified CD4+ T cells up to 3 days following IV cyclophosphamide 0.5 g/m2
  Other Names: cyclophosphamide
  Arms: Cohort 2 - IV cyclophosphamide 0.5 g/m2
Genetic: SB-728-T — Infusion will be 5 to 30 billion ZFN modified CD4+ T cells up to 3 days following IV cyclophosphamide 1.0 g/m2
  Other Names: cyclophosphamide
  Arms: Cohort 3 - IV cyclophosphamide 1.0 g/m2
Genetic: SB-728-T — Infusion will be 5 to 30 billion ZFN modified CD4+ T cells up to 3 days following IV cyclophosphamide 2.0 g/m2
  Other Names: cyclophosphamide
  Arms: Cohort 4 - IV cyclophosphamide 2.0 g/m2
Genetic: SB-728-T — Infusion will be 5 to 30 billion ZFN modified CD4+ T cells up to 3 days following IV cyclophosphamide 1.5 g/m2
  Other Names: cyclophosphamide
  Arms: Cohort 5 - IV cyclophosphamide 1.5 g/m2

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and effect on HIV viral load, of escalating doses of cyclophosphamide administered 1 day prior to SB-728-T infusion.

DETAILED DESCRIPTION:
The objectives of the study are to augment HIV-specific T-cells and to reverse or decrease the progressive destruction of CD4+ T-cells that leads to clinical AIDS. Levels of engraftment vary from negligible to about 10% of the CD4+ T-cells in the vascular compartment. Preliminary analyses of HAART TI suggest that an anti-HIV effect may correlate with the level of SB-728-T engraftment. Concurrently, non-myeloablative lymphodepletion with cyclophosphamide has been demonstrated to enhance engraftment of adoptively transferred T-cells through a variety of mechanisms. The study is being undertaken to increase SB-728-T engraftment through the administration of low non-myeloablative doses of cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older with documented HIV diagnosis within 10 years of screening.
* Must be willing to comply with study-mandated evaluations; including discontinuation of current antiretroviral therapy during the treatment interruption.
* Must have received at least 6 months of continuous HAART therapy and have had undetectable VLs for the preceding 3 months.
* On stable antiretroviral medication (no changes to treatment within 4 weeks of screening.
* CD4+ T-cell count ≥500 cells/µL.
* Undetectable HIV-1 RNA obtained at screening.
* ANC ≥2500/µL
* Platelet count ≥200,000/µL

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection.
* Active or recent (in prior 6 months) AIDS defining complication.
* Any cancer or malignancy within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin or low grade (0 or 1) anal or cervical dysplasia.
* Current diagnosis of NYHA grade 3 or 4 CHF, uncontrolled angina or arrhythmias.
* History or any features on physical examination indicative of a bleeding diathesis.
* Received HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector.
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents within 30 days prior to screening.
* Use of Aspirin, dipyridamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2 week period prior to leukapheresis.
* Currently participating in another clinical trial or participation in such a trial within 30 days prior to screening visit.
* Subjects who are currently taking maraviroc or have received maraviroc within 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - UCLA Care Center, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Circle CARE Center, LLC, Norwalk, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Central West Clinical Research, Inc., St Louis, Missouri
  - Southwest CARE Center, Santa Fe, New Mexico
  - Ricky K Hsu, MD, PC, New York, New York
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Gordon Crofoot, MD, PA, Houston, Texas
- Clinical Research Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
Started | 3 | 6 | 11 | 3 | 3
Completed | 3 | 4 | 11 | 3 | 3
Not Completed | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2 | Total
Number analyzed (Participants) | 3 | 6 | 11 | 3 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (8.08) | 43.2 (6.11) | 41.5 (12.13) | 35.3 (10.21) | 50.0 (1.00) | 42.5 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 0 | 2
  Male | 3 | 5 | 10 | 3 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 0 | 1 | 6
  Not Hispanic or Latino | 3 | 4 | 8 | 3 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 2 | 6 | 9 | 2 | 2 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: Number of Participants with Treatment related Adverse Events in subjects who received any portion of the SB-728-T infusion
Time Frame: 28 days after the SB-728-T infusion of the last subject in each Cohort and up to 12 months
Measure: Number; unit: participants
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
Number analyzed (Participants) | 3 | 6 | 11 | 3 | 3
participants | 3 | 6 | 11 | 3 | 3

2. Secondary Outcome: Effect of Escalating Doses of Cyclophosphamide on SB-728-T Engraftment as Measured by CCR5 Modified CD4 Cells in Blood.
Description: Effect of repeat doses of SB-728-T on engraftment following cyclophosphamide conditioning as measured by CCR5 Modified CD4 Cells in blood at Month 12.
Time Frame: Up to 12 months after the last SB-728-T infusion
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: cells 10^9/L
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
Number analyzed (Participants) | 3 | 4 | 10 | 3 | 3
cells 10^9/L | 0.038 (0.0409) | 0.061 (0.0447) | 0.143 (0.1055) | 0.085 (0.0197) | 0.079 (0.0155)

3. Secondary Outcome: Effect of SB-728-T on Plasma HIV-1 RNA Levels Following HAART Interruption
Description: Effect of SB-728-T on plasma HIV-1 RNA levels following HAART interruption. The unit is log copies/mL, except for the Cohort 1, the unit is " copies/mL".
  Cohort 1 mean and SD are 0. All 3 subjects had NO HIV-1 RNA DETECTED.
Time Frame: Up to 12 months after the last SB-728-T infusion
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: log copies/mL
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
Number analyzed (Participants) | 3 | 4 | 11 | 3 | 3
log copies/mL | 0 (0) | 0.250 (0.5000) | 1.537 (1.3955) | 0.667 (0.5774) | 3.442 (1.1545)

4. Secondary Outcome: Change From Baseline to Month 12 in CD4+ T-cell Counts in Peripheral Blood After Repeat Treatments With SB-728-T. (i.e. Month 12 Value - Baseline Value)
Description: Change from baseline to month 12 in CD4+ T-cell counts in peripheral blood after repeat treatments with SB-728-T. (i.e. month 12 value - baseline value)
Time Frame: Up to 12 months after the last SB-728-T infusion
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: cells 10^9/L
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
Number analyzed (Participants) | 3 | 4 | 10 | 3 | 3
cells 10^9/L | 0.064 (0.1309) | 0.149 (0.3736) | -0.043 (0.1712) | 0.153 (0.3247) | 0.099 (0.3279)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1 - IV Cyclophosphamide 200 mg | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 | Cohort 5 - IV Cyclophosphamide 1.5 g/m2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/11 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 0/11 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 11/11 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - IV Cyclophosphamide 200 mg (N=3) | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 (N=6) | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 (N=11) | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 (N=3) | Cohort 5 - IV Cyclophosphamide 1.5 g/m2 (N=3)
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - IV Cyclophosphamide 200 mg (N=3) | Cohort 2 - IV Cyclophosphamide 0.5 g/m2 (N=6) | Cohort 3 - IV Cyclophosphamide 1.0 g/m2 (N=11) | Cohort 4 - IV Cyclophosphamide 2.0 g/m2 (N=3) | Cohort 5 - IV Cyclophosphamide 1.5 g/m2 (N=3)
Nausea (Gastrointestinal disorders) | 2 | 4 | 4 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 4 | 3 | 3 | 0
Pyrexia (General disorders) | 1 | 2 | 6 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 3 | 0 | 2
Pain (General disorders) | 1 | 1 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 3 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 1 | 1
Furuncle (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Scintillating scotoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Syphilis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nervous system disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6 | 4 | 1 | 2
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 4 | 1 | 1
Migraine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Psychiatric disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 0
Agitation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Insomnia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Substance abuse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders (Renal and urinary disorders) | 0 | 1 | 4 | 1 | 1
Cough (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Sinus congestion (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Skin odour abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Pallor (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed written materials related to the study or an outline of any proposed oral presentations, shall be submitted to Sangamo for approval at least 45 days prior to submission of materials for publication or any oral disclosure to a third party. If Sangamo determines that a description of patentable subject matter is contained in such written material or outline, it shall notify the clinical site within 1 month after receipt and Sangamo will have an additional 90 days for review.

DOCUMENTS (2):
  • Study Protocol (2014-01-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT01543152/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT01543152/SAP_001.pdf